CLINICAL TRIAL: NCT01329796
Title: Pertubation With Lignocaine in Endometriosis Associated Symptoms Effect Study
Brief Title: Pertubation With Lignocaine in Endometriosis
Acronym: PLEASE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isifer AB (Industry)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Karin Wickström, Danderyd Hospital, Stockholm, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISI-06-01
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-04

CONDITIONS: Endometriosis; Dysmenorrhea
Keywords: dysmenorrhea,; pelvic pain; dyspareunia; endometriosis
MeSH Terms: conditions — Endometriosis; Dysmenorrhea; Pelvic Pain; Dyspareunia | interventions — Lidocaine; Ringer's Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pertubation with Endole® (lignocaine) (Experimental): Three treatments were to be given preovulatory at cycle day 6-12 in three sequential menstrual cycles.
  Interventions: Drug: Lignocaine
- Placebo (Placebo Comparator): Pertubation with Ringer solution, given preovulatory at cycle day 6-12 in three sequential menstrual cycles.
  Interventions: Drug: Ringers Solution

INTERVENTIONS:
Drug: Lignocaine — Intrauterine flushing, pertubation, three treatments given preovulatory at cycle day 6-12 in three sequential menstrual cycles.
  Other Names: Lidocaine
  Arms: Pertubation with Endole® (lignocaine)
Drug: Ringers Solution — Intrauterine flushing, pertubation, given preovulatory at cycle day 6-12 in three sequential menstrual cycles.
  Arms: Placebo

SUMMARY:
Endometriosis is a disease of unknown aetiology that can cause severe dysmenorrhea. An altered immune system with elevated levels of cytokines in the peritoneal fluid as well as increased density of nerve fibres, might explain the pathophysiology of dysmenorrhea in endometriosis patients. Lignocaine has anti-inflammatory properties and exerts effect on nerve endings and intra peritoneal macrophages. Pertubation with lignocaine might represent an alternative treatment for endometriosis related dysmenorrhea and avoids the side-effects related to hormonal treatments. A double blind randomized clinical trial, was carried out to evaluate pertubation with lignocaine as a therapy for dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20 years
* endometriosis verified by laparoscopy
* dysmenorrhea or pelvic pain defined as a pain-score of >50 mm (VAS)
* normal Fallopian tubes
* regular menstrual cycles 21-35 days
* treatment with oral contraceptives (OC) ongoing > 1 month and continued during the trial
* previous hormonal treatment discontinued > 1 month (OC, gestagens) and > 6 months (GnRH)
* no wish for pregnancy during the study
* normal Pap-smear
* negative Chlamydia-test
* negative pregnancy-test
* informed consent given and signed

Exclusion Criteria:

* Continuous treatment with medication that may increase risk for infection - clinical signs of pelvic inflammatory disease
* hyperreactivity to local anesthesia
* fibroids > 2 cm
* ongoing treatment with GnRH-analog
* ongoing continuous treatment with high dose gestagens
* pregnancy
* peritubal adhesions
* occluded Fallopian tubes
* inability to understand information or comply with the study procedures
* participation in a clinical study within one year before the present study
* any disease or laboratory finding considered of importance by the investigator not to include the patient

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-03; Primary Completion 2009-06 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Pain-questionnaire (validated for endometriosis) supplemented with VAS-scale. | After three pertubations
  The pain-questionnaire will be filled out: first time during the first period after inclusion in the study (1st menstruation prior to study treatments=baseline for evaluation) and thereafter during 2nd, 3rd, 4 th, 7th, 10th and 13th menstrual periods.

SECONDARY OUTCOMES:
Quality of life-questionnaire (validated), EHP-30 | At the 7th menstruation i.e. after approximately 6 months.
  The Quality of life-questionnaire will be filled out: first time during the first period after inclusion in the study (1st menstruation prior to study treatment=baseline for evaluation) and thereafter during 7th and 13th menstrual period.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Wickström, MD, Principal Investigator — Danderyd Hospital, SE-182 88 Stockholm, Sweden; Greta Edelstam, MD, Study Director — Karolinska University Hospital at Huddinge SE-141 86 Stockholm, Sweden
Locations (3):
- Sweden (3):
  - Läkargruppen Victoria Söderhallarna 120, Stockholm, Stockholm County
  - Karolinska Institute, Fertility Unit, K59 Karolinska University Hospital at Huddinge, Stockholm, Stockholm County
  - Department of Gynaecology and Obstetrics Danderyd Hospital, Stockholm, Stockholm County

REFERENCES:
- [Derived] Wickstrom K, Edelstam G. Minimal clinically important difference for pain on the VAS scale and the relation to quality of life in women with endometriosis. Sex Reprod Healthc. 2017 Oct;13:35-40. doi: 10.1016/j.srhc.2017.05.004. Epub 2017 May 25. PMID 28844356
- [Derived] Wickstrom K, Spira J, Edelstam G. Serum concentration of lignocaine after pertubation: an observational study. Drugs R D. 2013 Sep;13(3):235-9. doi: 10.1007/s40268-013-0022-8. PMID 23921822
- [Derived] Wickstrom K, Bruse C, Sjosten A, Spira J, Edelstam G. Pertubation with lignocaine as a new treatment of dysmenorrhea due to endometriosis: a randomized controlled trial. Hum Reprod. 2012 Mar;27(3):695-701. doi: 10.1093/humrep/der434. Epub 2012 Jan 9. PMID 22232129